CLINICAL TRIAL: NCT04361968
Title: Combining Animal-assisted Intervention and Placebo-induced Analgesia: The Dog as Treatment in a Randomized Controlled Trial
Brief Title: Combining Animal-assisted Intervention and Placebo-induced Analgesia
Acronym: AIPLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Dr. phil. Karin Hediger, Faculty of Psychology, University of Basel, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020- 00642
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Pain; Therapeutic Alliance; Placebo
Keywords: Treatment Rationale; animal-assisted intervention
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled parallel group within-subjects design
Who Masked: Participant
Masking Description: As the employed study design necessitates the deception of participants about the true nature of the used intervention, i.e. placebo cream and the true aim of the dog's presence.
  After the termination of the study, all the subjects are debriefed regarding the real experimental procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Animal-assisted placebo condition (Experimental): Participants receive verbal information that they are receiving an analgesic cream. Additionally, and before getting the dog, participants will get a therapeutic rationale for the presence of the dog.
  Interventions: Other: Animal-assisted placebo condition
- Placebo condition (Experimental): Participants receive verbal information that they are receiving an analgesic cream.
  Interventions: Other: Placebo condition
- Dog only condition (Experimental): Before meeting the dog, participants will get a therapeutic rationale for the presence of the dog.
  Interventions: Other: Dog only condition
- Control condition (Other): Participants in this condition will receive no intervention.
  Interventions: Other: Control Condition

INTERVENTIONS:
Other: Animal-assisted placebo condition — Participants receive the same verbal information as in the Placebo condition. Additionally, participants will receive the same verbal information as in the Dog only condition.
  Arms: Animal-assisted placebo condition
Other: Placebo condition — Participants receive verbal information that they are receiving an analgesic cream (i.e. ""Antidolor, containing Lidocain"), which has been shown to produce significant pain reduction in previous clinical trials. However, they will receive an inert cream.
  Arms: Placebo condition
Other: Dog only condition — Participants will get a therapeutic rationale for the presence of the dog. The rationale is supported in the literature and therefore not invented for the purpose of this study. Participants will be told that: "Studies have shown the presence of an animal can affect pain perception because the presence and the interaction with an animal can increase our Oxytocin level. Therefore, the investigators want to examine if the presence of a dog has an impact on your pain perception. While participants have to wait for the action time of the cream they are allowed to pet the dog. The intensity of interaction will be documented and be rated on a scale from 1-5 (1=very low degree of interaction, 5=very high degree of interaction). During the experiment the dog will be lying in the room with some distance to participants to avoid further physical interaction. The dog will always be lying at the same spot. Participants will still be able to see the dog.
  Arms: Dog only condition
Other: Control Condition — Participants in this condition will receive no intervention. All instructions will be conveyed in a standardized manner to ensure that the participant-experimenter relationship is comparable in terms of friendliness and attention across all four conditions.
  Arms: Control condition

SUMMARY:
An increased interest of animal-assisted interventions (AAI) can be observed within clinical practice, even though it is still not entirely clear how the presence of an animal contributes to the outcome of a treatment. One theory maintains that the mere presence of an animal influences the therapeutic alliance between therapist and client.

However, results from a recent study suggest that a relationship between patient and health-provider alone is not sufficient to influence treatment outcomes, but that a therapeutic rationale is needed and that verbal instructions and suggestions are highly important in shaping participants' treatment expectations.

To investigate this theory, this study will combine AAI with a placebo intervention, as placebo interventions offer the basic form of intervention working through relationship and expectancy.

The effects of the presence of a dog will be assessed with a standardized experimental heat pain paradigm (TSA-II) in a randomized controlled trial in healthy participants (N=128).

After a baseline measurements of heat pain threshold and tolerance, participants will be randomly assigned to one of the following four conditions: a) placebo intervention , no dog present, b) placebo intervention, dog present, c) no placebo intervention, no dog present and d) no placebo intervention, dog present.

The dog will be introduced after randomization. Expectancy will be induced by telling participants that the contact to an animal increases the oxytocin level, which has an non inflammatory effect.

The placebo intervention will be a deceptive cream which is said to helps against pain.

Afterwards, posttreatment measurements will be conducted and participants fill in questionnaires about their perceptions of the experimenter.

DETAILED DESCRIPTION:
A growing body of literature suggests that animal-assisted interventions (AAI) have important clinical effects on humans, e.g. decreased physiological stress, reduction of depression and anxiety symptoms and reduction in pain perception and experience. Such evidence leads to an increased interest in using AAI in clinical practice. However, it is still not quite clear how AAI works or in other words what it is that makes AAI effective. Therefore, it is crucial to investigate how the inclusion of animals in clinical practice contributes to beneficial therapeutic outcomes.

In this regard, it has been assumed that the presence of an animal enhances the development of the therapeutic alliance, which, in turn, has been shown to play a crucial role in the outcome of the treatment.

However, results from a recent study suggest that a relationship between patient and health-provider alone is not sufficient to influence treatment outcomes, but that a therapeutic rationale is needed and that verbal instructions and suggestions are highly important in shaping participants' treatment expectations.

As placebo effects are related to therapeutic rationale and relationship, the investigators would like to use an expectancy-induced placebo intervention to identify if animal-assisted intervention also works through these two components.

Given that placebo analgesia works well through therapeutic rationale the investigators decided to employ an animal-integrated placebo intervention study with healthy participants (N=128) in a standardized experimental heat pain paradigm. Even though a growing body of evidence highlights the positive effects of animal-assisted interventions until this day little is known about the mechanisms. There exist various hypotheses trying to explain why AAI works, most focusing on the crucial role of the animal in the intervention. However, to the best of the investigator's knowledge there has been no study which examined if the effectiveness of animal-assisted interventions could simply be explained by the power of the therapeutic rational and the relationship. Therefore, it is still unknown if AAI is effective because of the animal or because of its influence on the therapeutic relationship and the given therapeutic rationale.

It is important to understand how AAI works. Moreover, if AAI, like other interventions, is about expectation and relationship, this could have important implications for clinical practice and a better understanding of how AAI must be used to be effective.

If AAI works through similar mechanisms as the placebo, then both interventions should have a similar impact on the outcome of the intervention (reduced pain perception, increased placebo analgesia). Findings of this study could have important implications, not only for clinical practice of AAI but also for intervention in general as the results could help to better understand the importance of these two components.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Right-handedness

Exclusion Criteria:

* Being scared of dogs by self-report
* dog hair allergy by self-report
* Any acute or chronic disease (chronic pain, hypertension, heart disease, renal disease, liver disease, diabetes) as well as skin pathologies, neuropathies or nerve entrapment symptoms, sensory abnormalities affecting the tactile or thermal modality
* Pregnancy
* Current medications (psychoactive medication, narcotics, intake of analgesics) or being currently in psychological or psychiatric treatment
* Insufficient German language skills to understand the instructions
* Previous participation in studies using pain assessment with Peltier Devices
* Current or regular drug consumption (THC, cocaine, heroin, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Posttreatment objective heat pain tolerance | 10 minutes
  Heat stimuli will be administered to the right volar forearm using a 30x 30-mm Peltier device (Medoc, Ramatishai, Israel; TSA-II) placed at 2/3 of the distance from wrist to elbow. Pain tolerance will be determined by the method of limits: Participants will be asked to stop the increasing heat stimulus at the moment they cannot stand the heat any longer. Three measurements will start at 32 °C, with a rise of 0.5 °C/s. Heat tolerance will be defined as the average of the three measurements.
Corresponding subjective ratings of pain intensity and unpleasantness of pain tolerance | 5 minutes
  Subjective ratings of pain intensity and unpleasantness will be measured with a visual analogue scale (VAS): Following each pain stimuli with the TSA-II participants have to respond on a VAS how intense and unpleasant the pain is. The range of the scale is from 1-10 (1= not intense/unpleasant at all; 10= the most intense/unpleasant pain).

SECONDARY OUTCOMES:
Posttreatment objective heat threshold | 10 minutes
  Heat pain threshold will be determined by the methods of limits. Temperature will be increased from the baseline (32°C) at a rate of 0.5°C /s. Participants are instructed to press the button to determine the turning point from perceiving warmth to the perception of pain. When the pain threshold has been reached, the device will resume from its baseline (32 °C) with a rise of 0.5 °C/s. This procedure will be repeated three times. Pain threshold will be defined as the average of the three measurements.
Corresponding subjective ratings of pain intensity and unpleasantness of pain threshold. | 5 minutes
  Subjective ratings of pain intensity and unpleasantness will be measured with a visual analogue scale. ): Following each pain stimuli with the TSA-II participants have to respond on a VAS how intense and unpleasant the pain is. The range of the scale is from 1-10 (1= not intense/unpleasant at all; 10= the most intense/unpleasant pain).
Pain expectancy and relief | 2 minutes
  The Expectancy of Relief Scale assesses how intensive and unpleasantness participants expect the pain to be after the treatment phase. The expectancy ratings are made on the same VAS (ranging from 1 to 10, (1= not intense/unpleasant at all; 10= the most intense/unpleasant pain) as those for pain intensity and pain unpleasantness.
Participants perception of the study conductor assessed by questionnaire | 10 minutes
  Participants perception of the study conductor will be assessed with the Counselor Rating Form (CRF) Short questionnaire. The CRF-S assesses participant's perception of the study conductor and if their perception changes in the presence of absence of a dog. The CRF-S is a brief 12-items questionnaire that has been developed to measure people's perception of a therapist on total three subscales: trustworthiness, expertness and attractiveness (Corrigan and Schmidt, 1983). The questionnaire contains item such as "honest", "likeable", "trustworthy", "friendly" on a 7-point Likert scale ranging from 1 (not very) to 7 (very). This questionnaire will be used after baseline heat pain measurements and a second time after posttreatment heat pain measurements.
Attitude towards dogs assessed by questionnaire | 2 minutes
  Attitude towards dogs will be assessed with the questionnaire on the attitude towards dogs (AAPL). This questionnaire was designed for this study. This questionnaire assesses if participants like dogs and animals. This study developed this questionnaire for this study.
Kontextmodellfragebogen (KMF)/context model questionnaire | 5 minutes
  The KMF assesses the perception of participants of the study conductor and the credibility and expectation of the intervention. Participants fill out this questionnaire after the treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Hediger, Dr. phil, Study Chair — Clinical Psychology and Psychotherapy, University of Basel
Locations (1):
- Division of Clinical Psychology and Psychotherapy, University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
The investigators are planning on sharing the anonymized data on an openly assess platform.

REFERENCES:
- [Background] Kelley JM, Kraft-Todd G, Schapira L, Kossowsky J, Riess H. The influence of the patient-clinician relationship on healthcare outcomes: a systematic review and meta-analysis of randomized controlled trials. PLoS One. 2014 Apr 9;9(4):e94207. doi: 10.1371/journal.pone.0094207. eCollection 2014. PMID 24718585
- [Background] Birkhauer J, Gaab J, Kossowsky J, Hasler S, Krummenacher P, Werner C, Gerger H. Trust in the health care professional and health outcome: A meta-analysis. PLoS One. 2017 Feb 7;12(2):e0170988. doi: 10.1371/journal.pone.0170988. eCollection 2017. PMID 28170443
- [Background] Antonioli C, Reveley MA. Randomised controlled trial of animal facilitated therapy with dolphins in the treatment of depression. BMJ. 2005 Nov 26;331(7527):1231. doi: 10.1136/bmj.331.7527.1231. PMID 16308382
- [Background] Calcaterra V, Veggiotti P, Palestrini C, De Giorgis V, Raschetti R, Tumminelli M, Mencherini S, Papotti F, Klersy C, Albertini R, Ostuni S, Pelizzo G. Post-operative benefits of animal-assisted therapy in pediatric surgery: a randomised study. PLoS One. 2015 Jun 3;10(6):e0125813. doi: 10.1371/journal.pone.0125813. eCollection 2015. PMID 26039494
- [Background] Colloca L, Sigaudo M, Benedetti F. The role of learning in nocebo and placebo effects. Pain. 2008 May;136(1-2):211-8. doi: 10.1016/j.pain.2008.02.006. Epub 2008 Mar 26. PMID 18372113
- [Background] Creary, P. (2017). The influence of the presence of a dog or cat on perceptions of a psychotherapist.
- [Background] Fluckiger C, Del Re AC, Wampold BE, Symonds D, Horvath AO. How central is the alliance in psychotherapy? A multilevel longitudinal meta-analysis. J Couns Psychol. 2012 Jan;59(1):10-7. doi: 10.1037/a0025749. Epub 2011 Oct 10. PMID 21988681
- [Background] Waite TC, Hamilton L, O'Brien W. A meta-analysis of Animal Assisted Interventions targeting pain, anxiety and distress in medical settings. Complement Ther Clin Pract. 2018 Nov;33:49-55. doi: 10.1016/j.ctcp.2018.07.006. Epub 2018 Jul 20. PMID 30396626
- [Background] Vase L, Riley JL 3rd, Price DD. A comparison of placebo effects in clinical analgesic trials versus studies of placebo analgesia. Pain. 2002 Oct;99(3):443-452. doi: 10.1016/S0304-3959(02)00205-1. PMID 12406519
- [Background] Del Re AC, Fluckiger C, Horvath AO, Symonds D, Wampold BE. Therapist effects in the therapeutic alliance-outcome relationship: a restricted-maximum likelihood meta-analysis. Clin Psychol Rev. 2012 Nov;32(7):642-9. doi: 10.1016/j.cpr.2012.07.002. Epub 2012 Jul 21. PMID 22922705
- [Background] Ein N, Li L, Vickers K. The effect of pet therapy on the physiological and subjective stress response: A meta-analysis. Stress Health. 2018 Oct;34(4):477-489. doi: 10.1002/smi.2812. Epub 2018 Jun 8. PMID 29882342
- [Background] Fiori G, Marzi T, Bartoli F, Bruni C, Ciceroni C, Palomba M, Zolferino M, Corsi E, Galimberti M, Moggi Pignone A, Viggiano MP, Guiducci S, Calamai M, Matucci-Cerinic M. The challenge of pet therapy in systemic sclerosis: evidence for an impact on pain, anxiety, neuroticism and social interaction. Clin Exp Rheumatol. 2018 Jul-Aug;36 Suppl 113(4):135-141. Epub 2018 Sep 20. PMID 30277859
- [Background] Gaab J, Kossowsky J, Ehlert U, Locher C. Effects and Components of Placebos with a Psychological Treatment Rationale - Three Randomized-Controlled Studies. Sci Rep. 2019 Feb 5;9(1):1421. doi: 10.1038/s41598-018-37945-1. PMID 30723231
- [Background] Hsieh C, Kong J, Kirsch I, Edwards RR, Jensen KB, Kaptchuk TJ, Gollub RL. Well-loved music robustly relieves pain: a randomized, controlled trial. PLoS One. 2014 Sep 11;9(9):e107390. doi: 10.1371/journal.pone.0107390. eCollection 2014. PMID 25211164
- [Background] Kirsch I, Weixel LJ. Double-blind versus deceptive administration of a placebo. Behav Neurosci. 1988 Apr;102(2):319-23. doi: 10.1037//0735-7044.102.2.319. PMID 3365327
- [Background] Kruger, K. A. and J. A. Serpell (2010). Animal-assisted interventions in mental health: Definitions and theoretical foundations. Handbook on animal-assisted therapy, Elsevier: 33-48.
- [Background] Krummenacher P, Candia V, Folkers G, Schedlowski M, Schonbachler G. Prefrontal cortex modulates placebo analgesia. Pain. 2010 Mar;148(3):368-374. doi: 10.1016/j.pain.2009.09.033. Epub 2009 Oct 28. PMID 19875233
- [Background] Krummenacher P, Kossowsky J, Schwarz C, Brugger P, Kelley JM, Meyer A, Gaab J. Expectancy-induced placebo analgesia in children and the role of magical thinking. J Pain. 2014 Dec;15(12):1282-93. doi: 10.1016/j.jpain.2014.09.005. Epub 2014 Sep 23. PMID 25261340
- [Background] Le Roux, M. C. and R. Kemp (2009).
- [Background] Locher C, Frey Nascimento A, Kirsch I, Kossowsky J, Meyer A, Gaab J. Is the rationale more important than deception? A randomized controlled trial of open-label placebo analgesia. Pain. 2017 Dec;158(12):2320-2328. doi: 10.1097/j.pain.0000000000001012. PMID 28708766
- [Background] Odendaal JS. Animal-assisted therapy - magic or medicine? J Psychosom Res. 2000 Oct;49(4):275-80. doi: 10.1016/s0022-3999(00)00183-5. PMID 11119784
- [Background] Odendaal JS, Meintjes RA. Neurophysiological correlates of affiliative behaviour between humans and dogs. Vet J. 2003 May;165(3):296-301. doi: 10.1016/s1090-0233(02)00237-x. PMID 12672376
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Petersson M, Alster P, Lundeberg T, Uvnas-Moberg K. Oxytocin increases nociceptive thresholds in a long-term perspective in female and male rats. Neurosci Lett. 1996 Jul 12;212(2):87-90. doi: 10.1016/0304-3940(96)12773-7. PMID 8832645
- [Background] Petersson M, Eklund M, Uvnas-Moberg K. Oxytocin decreases corticosterone and nociception and increases motor activity in OVX rats. Maturitas. 2005 Aug 16;51(4):426-33. doi: 10.1016/j.maturitas.2004.10.005. Epub 2004 Dec 25. PMID 16039417
- [Background] Petrovic P, Dietrich T, Fransson P, Andersson J, Carlsson K, Ingvar M. Placebo in emotional processing--induced expectations of anxiety relief activate a generalized modulatory network. Neuron. 2005 Jun 16;46(6):957-69. doi: 10.1016/j.neuron.2005.05.023. PMID 15953423
- [Background] Pollo A, Amanzio M, Arslanian A, Casadio C, Maggi G, Benedetti F. Response expectancies in placebo analgesia and their clinical relevance. Pain. 2001 Jul;93(1):77-84. doi: 10.1016/S0304-3959(01)00296-2. PMID 11406341
- [Background] Souter, M. A. and M. D. Miller (2007).
- [Background] Corrigan, J. D., & Schmidt, L. D. (1983). Development and validation of revisions in the Counselor Rating Form. Journal of Counseling Psychology, 30(1), 64.
- [Background] Horvath AO, Del Re AC, Fluckiger C, Symonds D. Alliance in individual psychotherapy. Psychotherapy (Chic). 2011 Mar;48(1):9-16. doi: 10.1037/a0022186. PMID 21401269
- [Background] Hoffmann, A. O., et al. (2009).
- [Derived] Wagner C, Gaab J, Hediger K. The Importance of the Treatment Rationale for Pain in Animal-Assisted Interventions: A Randomized Controlled Trial in Healthy Participants. J Pain. 2023 Jun;24(6):1080-1093. doi: 10.1016/j.jpain.2023.01.004. Epub 2023 Jan 12. PMID 36641027